CLINICAL TRIAL: NCT05266495
Title: Effectiveness of Brolucizumab in Pretreated Patients With nAMD in the Real-world Setting in Gulf Countries United Arab of Emirates, Kuwait , Bahrain , Oman and Qatar
Brief Title: Effectiveness of Brolucizumab in Pre-treated Patients With nAMD in the Real-world Setting
Status: Terminated | Type: Observational
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AAE01
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-03

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD; brolucizumab; NIS
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brolucizumab: patients who received their first injection of Brolucizumab either during the active recruitment period (1 year prospective) or during the 6 months pre-start of the recruitment (6 months retrospective)
  Interventions: Other: Brolucizumab

INTERVENTIONS:
Other: Brolucizumab — There is no treatment allocation. Patients administered brolucizumab by prescription will be enrolled.

SUMMARY:
The study is a prospective and retrospective, observational, single-arm, non-randomized cohort study of ocular treatment with intravitreal injections of brolucizumab in nAMD patients. This study will be conducted prospectively and retrospectively (for patients who had their first brolucizumab injection before study start) using data collected in a standardized manner.

DETAILED DESCRIPTION:
Retrospective data will be collected for all patients starting treatment with brolucizumab for up to 12 months before baseline.

Patients who received brolucizumab before the study start will be recruited into the study and presented an informed consent form (ICF) at their first visit. Their index date will be the date of their first brolucizumab injection, which must have occurred during the recruitment period or in 6 months prior to the first visit in the recruitment period. Patient history and characteristics will be recorded in the 12 months prior to the index date.

Index date (Baseline): defined as the date of the first anti-VEGF injection (brolucizumab) in the patient study eye.

Index period: The patients fulfilling the inclusion criteria will be identified during the period 01-Nov-2021 and onwards.

Study period: The period is between May-2020 and Nov-2023 to allow 6-month pre-index period and at least a 12-month follow-up period for each recruited patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nAMD
* Patients with ≥18 years of age at index
* Receipt of at least one injection of brolucizumab (not necessarily the first one) during the index period
* Signed informed consent

Exclusion Criteria:

* Patients treated for retinal vein occlusion (RVO), diabetic macular edema (DME), myopic choroidal neovascularization (mCNV), and have diagnoses of diabetes-related macular degeneration within 6 months prior to the index date
* Receipt of any anti-VEGF treatment other than brolucizumab in the study eye during the index period
* Receipt of brolucizumab in the study eye more than 6 months before the index period, i.e., brolucizumab treatment started more than 6 months before the start of the study
* Any active intraocular or periocular infection or active intraocular inflammation in the study eye at index date
* Patients who have any contraindication and are not eligible for treatment with brolucizumab as according to the label
* Patients who were treated with more than 2 types of anti-VEGF before index date (4th line brolucizumab patients or more)
* Any medical or psychological condition in the treating physician's opinion which may prevent the patient from the 12-month study participation
* Patients participating in parallel in an interventional clinical trial Note: if a patient experiences an adverse event (AE), they may still be recruited in another study following this AE if they fulfill their inclusion criteria. Their data will still be collected as planned by the current protocol
* Patients participating in parallel in any other NIS generating primary data for an anti-VEGF drug

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that started brolucizumab treatment during the study recruitment period or patients that started brolucizumab treatment during the 6 months preceding the start of study recruitment
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with absence of SRF and IRF | Month 12
  percentage of treated patients with absence of SRF and IRF. Patients who have discontinued brolucizumab before Month 12 will be counted as not having achieved the endpoint of fluid resolution (absence of SRF and IRF), unless they reached it at the last visit while still on brolucizumab treatment before the discontinuation.

SECONDARY OUTCOMES:
Percentage of patients ≥ 80 years old | Baseline
  Percentage of patients ≥ 80 years old will be collected
Duration of diagnosis | Baseline
  Time since first diagnosis (years) will be collected
Percentage of patients with baseline visit | Baseline
  Percentage of patients with baseline visit will be collected
Percentage of patients with bilateral disease | Baseline
  Percentage of patients with bilateral disease will be collected
Percentage of patients with lesion type | Baseline
  Percentage of patients by lesion type will be collected: occult, minimally classic, predominantly classic, other
Percentage of patients with presence of SRF, IRF and sub-RPE | Baseline
  It will be collected the percentage of patients with presence of:
  * Subretinal Fluid (SRF)
  * Intra-Retinal Fluid (IRF)
  * Subretinal Fluid (SRF) and/or Intra-Retinal Fluid (IRF)
  * Sub-Retinal Pigment Epithelium
Baseline CST | Baseline, Month 3, Month 6, Month 9 and Month 12
  Central Subfield Thickness (CST) in μm will be collected
Baseline VA | Baseline
  Visual Acuity (VA) will be measured with Early Treatment Diabetic Retinopathy Study (ETDRS) letters.
  Conversion of VA readings to approximate ETDRS Letters:
  For Snellen fraction decimal >0.025 (< logMAR1.60) the following formula is used: approximate ETDRS letters = 85+50*log10(Snellen fraction)
  For Snellen fractions decimal ≤ 0.025 four bins are defined:
  * > 0.020 to 0.025 (logMAR 1.70 to 1.60) is 5 letters
  * > 0.015 to 0.020 (logMAR 1.82 to 1.70) is 3 letters
  * > 0.005 to 0.015 (logMAR 2.30 to 1.82) is 1 letter
  * ≤ 0.005 (logMAR ≥ 2.30) is 0 letter
Percentage of patients with the study eye that has VA equal or less than the VA in fellow eye | Baseline
  Percentage of patients with the study eye that has Visual Acuity (VA) equal or less than the VA in fellow eye will be collected
Percentage of patients with baseline VA in the following categories (≤35, 36-69, ≥ 70 ETDRS letters) | Baseline
  Percentage of patients with baseline Visual Acuity (VA) in the following categories (≤35, 36-69, ≥ 70 ETDRS letters) will be collected
Percentage of patients with VA between 34 and 72 ETDRS letters | Baseline
  Percentage of patients with Visual Acuity (VA) within these values will be collected: 33 < VA < 73
Percentage of patients with baseline VA < 73 ETDRS letters and active (SRF only) | Baseline
  Percentage of patients with baseline VA < 73 ETDRS letters and active (SRF only) Active SRF is described as patients with new presence of SRF or increased SRF
Percentage of patients with different ethnic groups | Baseline
  Percentage of patients by ethnicity will be presented
Switch Patients: Previous anti-VEGF treatments of nAMD pre-treated patients | Baseline
  Previous anti-VEGF treatments of nAMD pre-treated patients will be collected
Switch Patients: Duration of previous anti-VEGF treatments | Baseline
  Duration of previous anti-VEGF treatments will be collected
Switch Patients: Number of injections in the last year before switching to brolucizumab | Baseline
  Number of injections in the last year before switching to brolucizumab will be collected
Switch Patients: Last interval of anti-VEGF treatment before switching | Baseline
  Last interval of anti-VEGF treatment before switching will be collected
Percentage of patients with absence of SRF | Month 3, Month 6, Month 9 and Month 12
  The total percentage of patients with absence of Subretinal Fluid (SRF) and percentage of patients with absence of SRF from those with presence of SRF at baseline will be collected
Percentage of patients with stable SRF | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with stable Subretinal Fluid (SRF), from those with absence of SRF at baseline
Time to absence of SRF during the 12-month treatment with brolucizumab | 12 months
  Time to absence of Subretinal Fluid (SRF) will be collected
Percentage of patients with absence of IRF | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with absence of Intra-Retinal Fluid (IRF), and percentage of patients with absence of IRF from those with presence of IRF at baseline will be collected
Percentage of patients with stable IRF | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with stable Intra-Retinal Fluid (IRF), from those with absence of IRF at baseline
Time to absence of IRF during the 12-month treatment with brolucizumab | 12 months
  Time to absence of Intra-Retinal Fluid (IRF) during the 12-month treatment with brolucizumab will be collected
Percentage of patients with absence of sub-RPE | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with absence of sub-Retinal Pigment Epithelium (RPE) and percentage of patients with absence of sub-RPE, from those with presence of sub-RPE at baseline will be collected
Percentage of patients with stable sub-RPE | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with stable sub-Retinal Pigment Epithelium (RPE), from those with absence of sub-RPE at baseline
Time to absence of sub-RPE during the 12-month treatment with brolucizumab | 12 months
  Time to absence of sub-Retinal Pigment Epithelium (RPE) during the 12-month treatment with brolucizumab will be collected
Percentage of patients with absence of SRF, IRF and sub-RPE | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with absence of Subretinal Fluid (SRF), Intra-Retinal Fluid (IRF) and sub-Retinal Pigment Epithelium (RPE) and percentage of patients with absence of SRF and IRF and sub-RPE, from those with presence of SRF or IRF or sub-RPE at baseline will be collected
Time to absence of IRF and SRF and sub-RPE during the 12-month treatment with brolucizumab | 12 months
  Time to absence of IRF and SRF and sub-RPE during the 12-month treatment with brolucizumab
Estimate CST change from baseline | Month 3, Month 6, Month 9 and Month 12
  Estimate Central Subfield Thickness (CST) change from baseline (in μm) will be collected
Percentage of patients with reduced CST vs baseline | Baseline, Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with reduced CST vs baseline will be collected
Association between CST variability at Months 1-12 and VA change from baseline | Month 3, Month 6, Month 9 and Month 12
  Correlation statistical tests between CST variability at Months 1-12 (quartiles) and VA change from baseline to Months 3, 6, 9 and 12
Association between CST variability at Months 1-12 and number of injections | Month 12
  Correlation statistical tests between CST variability at Months 1-12 (quartiles) and number of injections during the 12-month treatment with brolucizumab
Percentage of patients with clinician-graded subretinal fibrosis and/or macular atrophy | Month 12
  Percentage of patients with clinician-graded subretinal fibrosis and/or macular atrophy
VA change from baseline | Baseline, Month 3, Month 6, Month 9 and Month 12
  Visual Acuity (VA) change from baseline (in ETDRS letters)
Percentage of patients with VA change from baseline | Baseline, Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with Visual Acuity (VA) change from baseline categorized as: ≤ -20, ≤ -15, (-15, -10], (-10, -5], (-5, 5), [5, 10), [10, 15), ≥ 15, ≥ 20 (in ETDRS letters)
Percentage of patients with ≥ 70 ETDRS letters | Month 3, Month 6, Month 9 and Month 12
  Percentage of patients with ≥ 70 ETDRS letters will be collected
Number of brolucizumab visits | Over Months 1-3, 3-6, 6-12 and 1-12
  Number of brolucizumab injections, non-injection visits and total number of visits will be collected
Distribution of injection intervals | During Months 1-6 and 1-12
  Distribution of injection intervals < 4; [4, 6); [6, 8); [8, 10); [10, 12); ≥12 weeks will be collected
Percentage of patients with at least one duration of interval between injections | 12 months
  Percentage of patients with at least one duration of interval between injections < 4; [4, 6); [6, 8); [8, 10); [10, 12); ≥ 12 weeks (the maximum injection interval will be kept) One duration of interval is defined as the time between one injection and the following one
Percentage of patients with at least two consecutive duration of intervals between injections | 12 months
  Percentage of patients with at least two consecutive duration of intervals between injections < 4; [4, 6); [6, 8); [8, 10); [10, 12); ≥12 weeks (the maximum duration will be kept) Two consecutive duration of intervals is the time between one injection and the second consecutive one.
Percentage of switch patients from other anti-VEGF that prolonged injection intervals with brolucizumab | Month 6, Month 9 and Month 12
  Percentage of switch patients from other anti-VEGF that prolonged injection intervals with brolucizumab will be collected
Percentage of patients with ≥ 3 brolucizumab injections | Month 3
  Percentage of patients with ≥ 3 brolucizumab injections will be collected
Number of participants by last recorded injection interval | Month 6 and Month 12
  Number of participants by last recorded injection interval (in weeks)
Time between two consecutive brolucizumab injections | Over Months 1-3
  Time (in days) between two consecutive brolucizumab injections will be collected
Number of visits with/without OCT | Over Months 1-6 and 1-12
  Number of visits with/without Optical Coherence Tomography (OCT) will be collected
Association between number of OCT and CNV activity | Month 6, Month 9 and Month 12
  Correlation statistical tests between number of Optical Coherence Tomography (OCT) (0-1, 2-3, ≥ 4) and Choroidal Neovascularization (CNV) activity [active, active (SRF only), inactive]
Association between number of OCT and VA change from baseline | Month 6, Month 9 and Month 12
  Correlation statistical tests between number of Optical Coherence Tomography (OCT) (0-1, 2-3, ≥ 4) and Visual Acuity (VA) change from baseline (in ETDRS letters)
Association between number of OCT and number of injections | 12 months
  Correlation statistical tests between number of Optical Coherence Tomography (OCT) (0-1, 2-3, ≥ 4) at Months 6, 9 and 12 and number of injections during the Months 1-6, 1-9 and 1-12 of treatment with brolucizumab
proportion of participants by baseline CNV activity | Baseline
  Baseline Choroidal Neovascularization (CNV) activity (active, active (SRF only), inactive) will be collected
Proportion of participants with and without Loading phase | 12 months
  Proportion of participants with and without Loading phase will be collected. Loading phase (yes/no) defined as ≥ 3-injections within 90 days post-index
VA at the end of the loading phase | Month 3
  Visual Acuity (VA) at the end of the loading phase will be collected. Loading phase is defined as ≥ 3-injections within 90 days post-index
CNV activity at the end of the loading phase | Month 3
  Choroidal Neovascularization (CNV) activity at the end of the loading phase (active, active (SRF only), inactive) will be measured.
  Loading phase is defined as ≥ 3-injections within 90 days post-index
Number of injections during the maintenance phase | Over months 3-12
  Number of injections during the maintenance phase will me measured
Percentage of patients with geographic atrophy | 12 Months
  Percentage of patients with geographic atrophy will be measured
Percentage of patients with subretinal fibrosis | 12 Months
  Percentage of patients with subretinal fibrosis will be measured
Assessment of criteria for no retreatment | 12 months
  Percentage of patients by criteria for no retreatment will be measured. ( i.e., disease activity assessed by: VA, anatomic parameters, predetermined by regimen, other (e.g., organizational, patient choice, etc.)
Percentage of patients who switch to another anti-VEGF | 6 Months, 9 Months and 12 Months
  Percentage of patients who switch to another anti-VEGF during the first 6, 9 and 12 months of treatment with brolucizumab will be measured
VA at time of switch | Up to 12 months
  Visual Acuity (VA) at time of switch will be measured with Early Treatment Diabetic Retinopathy Study (ETDRS) letters.
Percentage of patients with activity at time of switch | Up to 12 months
  Percentage of patients with activity at time of switch:
  * Intra-Retinal Fluid (IRF) activity
  * Subretinal Fluid (SRF) activity
  * sub-Retinal Pigment Epithelium (RPE) activity
  * Central Subfield Thickness (CST) activity
  * Choroidal Neovascularization (CNV) activity
Percentage of switchers with full loading phase | 12 months
  Percentage of switchers with full loading phase will be collected Loading phase (yes/no) defined as ≥ 3-injections within 90 days post-index
Percentage of patients by injection rate at pre-switch period | Up to 12 months
  Percentage of patients by injection rate at pre-switch period will be collected
Reason for switching to another anti-VEGF | 12 months
  Percentage of patients by reason for switching to another anti-VEGF will be collected
Last recorded injection interval before switching | Month 6 and Month 12
  Last recorded injection interval (in weeks) before switching will be collected
Duration of brolucizumab treatment before switching | Up to month 12
  Duration of brolucizumab treatment before switching will be collected
Percentage of patients who discontinue therapy | Up to 12 months
  Percentage of patients who discontinue therapy and reasons for discontinuation. Discontinuation is defined as if anti-VEGF brolucizumab was stopped (including treatment switch to another anti-VEGF) at some point and never re-introduced for at least 180 days, while the patient has at least one clinical or anatomical assessment during that period
Days of persistence | Up to 12 Months
  Persistence is defined as the time (in days) on drug from from the initiation of anti-VEGF therapy with brolucizumab to its discontinuation (defined as injection gap of >180 days)
Percentage of patients with AEs | 12 Months
  Percentage of patients with AEs will be collected
AE rate | Month 3, Month 6, Month 9 and Month 12
  AE rate (per 10,000 injections) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258AAE01 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18151